CLINICAL TRIAL: NCT06046209
Title: Comparing Clariti Elite Versus Proclear 1 Day
Brief Title: Comparing a Monthly Replacement Lens Versus a Daily Disposable Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-23-36
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-01

CONDITIONS: Myopia
Keywords: Refractive Errors; Eye Diseases
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lens, then Test Lens (Experimental): Participants wore the Control Lens for 90 minutes, then the Test Lens for 90 minutes.
  Interventions: Device: Control Lens; Device: Test Lens
- Test Lens, then Control Lens (Experimental): Participants wore the Test Lens for 90 minutes, then the Control Lens for 90 minutes.
  Interventions: Device: Control Lens; Device: Test Lens

INTERVENTIONS:
Device: Control Lens — Daily disposable contact lens for 90 minutes
Device: Test Lens — Monthly replacement contact lens for 90 minutes

SUMMARY:
The purpose of this study was to compare subjective ratings of lens handling at insertion for a monthly replacement lens versus a daily disposable lens in habitual soft lens wearers.

DETAILED DESCRIPTION:
This was a non-dispensing, randomized, double-masked, crossover study. Participants wore 2 different contact lenses bilaterally over 4 study visits, all conducted on the same day. Estimated duration of involvement for each participant was 4 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Were 17 to 40 years of age and have full legal capacity to volunteer;
2. Had read and signed an information consent letter;
3. Were willing and able to follow instructions and maintain the appointment schedule;
4. Were habitual daily wearers of spherical single vision soft contact lenses to correct for distance vision in each eye
5. Were correctable to a visual acuity of 20/20 or better (in each eye) with sphero-cylindrical subjective refraction;
6. Had an astigmatism of ≤ 0.75DC in subjective refraction;
7. Could be fit with the study contact lenses with a power between -1.00 and -6.00DS; this translates to best corrected vision sphere refraction that vertexes to a CL power between -1.00 and -6.00 (inclusive) at screening visit.
8. Demonstrated an acceptable fit with the study lenses.

Exclusion Criteria:

1. Had taken part in another clinical research study within the last 14 days;
2. Were currently habitual wearers of toric, multifocal or monovision lenses.
3. Had worn any rigid contact lenses in the past 6 months
4. Were an extended lens wearer (i.e., sleeping with their lenses)
5. Had a difference of ≥1.5 D in best vision sphere subjective refraction between eyes;
6. Had amblyopia and/or distance strabismus/binocular vision problem;
7. Had any known active ocular disease, allergies and/or infection;
8. Had a systemic condition that in the opinion of the investigator may affect a study outcome variable;
9. Were using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
10. Had a known sensitivity to the diagnostic pharmaceuticals to be used in the study;
11. Had undergone refractive error surgery or intraocular surgery;
12. Were a member of CORE directly involved in the study.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Centre for Ocular Research and Education (CORE)
Locations (1):
- University of Waterloo School of Optometry & Vision Science, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Lens, Then Test Lens: Participants wore the Control Lens for 90 minutes (Period 1), and then the Test Lens for 90 minutes (Period 2)
- Test Lens, Then Control Lens: Participants wore the Test Lens for 90 minutes (Period 1), and then the Control Lens for 90 minutes (Period 2)
Period: Period 1: First Intervention-90 Minutes
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2: Second Intervention-90 Minutes
Arm/Group | Control Lens, Then Test Lens | Test Lens, Then Control Lens
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who were dispensed lenses and successfully completed the study
Arm/Group | Overall Study
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling at Insertion
Description: Participants completed subjective ratings of the ease of application of the study lenses to eye immediately after lens application on a 0-100 integer scale, where 100=very easy and 0=very difficult.
Time Frame: Immediately after lens application
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Lens: Participants that received Control lens during either the first or second period of the study.
- Test Lens: Participants that received Test lens during either the first or second period of the study.
Arm/Group | Control Lens | Test Lens
Number analyzed (Participants) | 30 | 30
score on a scale | 83 (16) | 93 (9)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 4 hours
Arm/Group | Control Lens | Test Lens
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT06046209/Prot_SAP_000.pdf